CLINICAL TRIAL: NCT05690191
Title: A Multicenter, Prospective, Observational Clinical Protocol for Chidamide in Combination With Rituximab and Lenalidomide (cR2) in Real-world Practice in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: Chidamide in Patients With Recurrent and Refractory Diffuse Large b
Status: Enrolling by invitation | Type: Observational
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: JD-LK-2021-095-02
Record Dates: First submitted 2022-12-05; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Lenalidomide; Rituximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chidamide in combination with rituximab and lenalidomide: Chidamide tablets: 20mg orally, twice a week (at least 3 days between doses); Rituximab injection: 375mg/m2 intravenously, once every 4 weeks (Q4w), on the first day of each cycle; Lenalidomide capsule: 25mg orally, once before going to bed every night, from day 1 to day 21 of each cycle
  Interventions: Drug: Chidamide; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Chidamide — Chidamide tablets: 20mg orally, twice a week (at least 3 days between doses
Drug: Lenalidomide — Lenalidomide capsule: 25mg orally, once before going to bed every night, from day 1 to day 21 of each cycle
Drug: Rituximab — Rituximab injection: 375mg/m2 intravenously, once every 4 weeks (Q4w), on the first day of each cycle

SUMMARY:
A Multicenter, Prospective, Observational Clinical Protocol for Chidamide in Combination With Rituximab and Lenalidomide (cR2) in Real-world Practice in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational investigator-initiated clinical study. The subjects were adults (18 years of age and older) diagnosed with relapsed/refractory diffuse large B-cell lymphoma who will begin cR2 therapy at the time of enrollment. Patients were required to complete a visit every 4 weeks, lasting 24 weeks from the first dosing of the study protocol. The first visit was considered an enrollment visit. The specific dosage of cR2 will be determined according to the standard clinical practice of the treating physician. Participation in the study did not affect treatment decisions. Patients who could not continue with the cR2 regimen would terminate the visit early and then withdraw from the study. According to the data collected from the experiment, the safety and effectiveness of the research scheme were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. The decision of treating physicians to make cR2 regimen was not related to whether they participated in the study or not;
2. Age 18 and above, no gender limitation;
3. Patients with pathologically confirmed diffuse large B-cell lymphoma (DLBCL) who have relapsed or failed to respond to at least one systemic therapy;
4. Have at least one measurable lesion: any length of lymph node lesion ≥1.5cm or any length of extrinsic lesion > 1cm;
5. The serum pregnancy test of female subjects of childbearing age was negative;
6. Understand the test procedure and content, and sign the informed consent voluntarily.

Exclusion Criteria:

1. The decision of treating physicians to make cR2 regimen was not related to whether they participated in the study or not;
2. Age 18 and above, no gender limitation;
3. Patients with pathologically confirmed diffuse large B-cell lymphoma (DLBCL) who have relapsed or failed to respond to at least one systemic therapy;
4. Have at least one measurable lesion: any length of lymph node lesion ≥1.5cm or any length of extrinsic lesion > 1cm;
5. The serum pregnancy test of female subjects of childbearing age was negative;
6. Understand the test procedure and content, and sign the informed consent voluntarily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diffuse Large B-cell Lymphoma
Sampling Method: Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 30 months
  Objective response rates assessed by the investigator

SECONDARY OUTCOMES:
Adverse Events | 30 months
  Incidence of adverse events

OTHER OUTCOMES:
Complete response rate | 30 months
  Complete response rate
Progression-free survival | 30 months
  Progression-free survival
Overall survival time | 30 months
  Overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Bingzong LI, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China